CLINICAL TRIAL: NCT07144566
Title: Implementation of a Nurse-Led Clinical Program to Decrease Sexual Dysfunction Among Gynecological Cancer Patient
Brief Title: Improving Sexual Health in Gynecological Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Leah Spiro, Clinical Research Nurse Scientist, Nurse Practitioner, Brawerman Nursing Institute, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 00004279
Record Dates: First submitted 2025-08-17; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Gynaecologic Cancer
Keywords: Survivorship; Sexual Health; Sexual Dysfunction; Gynecologic Cancer
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Sex Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nurse Led Sexual Health Intervention (Experimental): Gynecologic Cancer patients ages 30-65yo who completed treatment within 12 months will be offered a sexual health nurse led intervention during follow up visits to include a pelvic exam, focused sexual health assessment, sexual health plan of care, sexual health education, and specialty referrals as needed.
  Interventions: Other: Nurse Led Sexual Health Clinical Program Intervention

INTERVENTIONS:
Other: Nurse Led Sexual Health Clinical Program Intervention — In person visit with Advanced Practice Provider (APP) whom is an Advanced Practice Nurse Practitioner in Oncology. Visit will include a focused pelvic exam, sexual health treatment plan, sexual health education, and referrals that follow the current Sexual Health Survivorship NCCN guidelines. A post visit telephone will be provided by the APP 8 weeks after APP visit for follow up questions and further education if needed.
  Other Names: Sexual health education; Sexual health treatment plan; Sexual Health Referrals; Sexual health focused pelvic exam

SUMMARY:
The goal of this clinical trial is to test whether a nurse-led program can improve screening and referral rates for sexual dysfunction and improve sexual health care in individuals with gynecological cancer. The main questions it aims to answer are:

Does participation in a nurse-led program improve the treatment of sexual dysfunction in individuals with gynecological cancer?

Does the program increase the frequency of screenings and referrals for sexual dysfunction?

Participants will:

Complete a visit with an advanced practice provider.

Fill out the Female Sexual Function Index survey.

Allow the research team to review medical records.

ELIGIBILITY:
Inclusion:

* Patients with a gynecologic cancer history
* Patients ages 30-65 years old
* Patients must have completed cancer treatment within the past 12 months
* Patients may be on maintenance therapy

Exclusion:

* Any records flagged "break the glass" or "research opt-out."
* Patients with severe psychiatric disorders that would impair consent or participation
* Patients with neurological disorders affecting sexual function
* Patients with a history of sexual violence or sexual assault

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female born
Enrollment: 35 (Estimated)
Dates: Start 2025-09-02 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the nurse led clinical sexual health dysfunction program | 12 weeks
  Assess improvement in sexual dysfunction in gynecologic cancer survivors via the Female Sexual Function Index (FSFI).
Effectiveness of the nurse led clinical sexual health dysfunction program | 12 weeks
  Assess effectiveness of the nurse led clinical sexual dysfunction program via number of referrals and treatments in the chart before and after the intervention in gynecologic cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Leah Spiro, DNP, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Birch K, Chung S, Zion SR, MacEwan JP, Malecki MJ. Incremental Health Care Costs of Anxiety and Depression Among Medicare Beneficiaries With Cancer. JCO Oncol Pract. 2023 May;19(5):e660-e671. doi: 10.1200/OP.22.00555. Epub 2023 Feb 17. PMID 36800552
- [Result] Sitlinger A, Zafar SY. Health-Related Quality of Life: The Impact on Morbidity and Mortality. Surg Oncol Clin N Am. 2018 Oct;27(4):675-684. doi: 10.1016/j.soc.2018.05.008. Epub 2018 Jul 21. PMID 30213412
- [Result] Hungr C, Recklitis CJ, Wright AA, Bober SL. How does a single session group intervention improve sexual function in ovarian cancer survivors? A secondary analysis of effects of self-efficacy, knowledge and emotional distress. Psychol Health Med. 2020 Jan;25(1):110-120. doi: 10.1080/13548506.2019.1626452. Epub 2019 Jun 5. PMID 31167551
- [Result] Wang X, Wang N, Zhong L, Wang S, Zheng Y, Yang B, Zhang J, Lin Y, Wang Z. Prognostic value of depression and anxiety on breast cancer recurrence and mortality: a systematic review and meta-analysis of 282,203 patients. Mol Psychiatry. 2020 Dec;25(12):3186-3197. doi: 10.1038/s41380-020-00865-6. Epub 2020 Aug 20. PMID 32820237
- [Result] Seaborne LA, Peterson M, Kushner DM, Sobecki J, Rash JK. Development, Implementation, and Patient Perspectives of the Women's Integrative Sexual Health Program: A Program Designed to Address the Sexual Side Effects of Cancer Treatment. J Adv Pract Oncol. 2021 Jan-Feb;12(1):32-38. doi: 10.6004/jadpro.2021.12.1.3. Epub 2021 Jan 1. PMID 33552660
- [Result] Chow KM, Chan Yip WHC, Porter-Steele J, Siu KY, Choi KC. Nurse-led sexual rehabilitation to rebuild sexuality and intimacy after treatment for gynaecological cancer: a randomised controlled trial (abridged secondary publication). Hong Kong Med J. 2023 Aug;29 Suppl 4(4):26-30. No abstract available. PMID 37690804
- [Result] Sousa Rodrigues Guedes T, Barbosa Otoni Goncalves Guedes M, de Castro Santana R, Costa da Silva JF, Almeida Gomes Dantas A, Ochandorena-Acha M, Terradas-Monllor M, Jerez-Roig J, Bezerra de Souza DL. Sexual Dysfunction in Women with Cancer: A Systematic Review of Longitudinal Studies. Int J Environ Res Public Health. 2022 Sep 21;19(19):11921. doi: 10.3390/ijerph191911921. PMID 36231221
- [Result] Kaufman R, Agrawal L, Teplinsky E, Kiel L, Abioye O, Florez N. From diagnosis to survivorship addressing the sexuality of women during cancer. Oncologist. 2024 Dec 6;29(12):1014-1023. doi: 10.1093/oncolo/oyae242. PMID 39269314

DOCUMENTS (2):
  • Study Protocol (2025-07-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT07144566/Prot_000.pdf
  • Informed Consent Form (2025-08-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT07144566/ICF_001.pdf